CLINICAL TRIAL: NCT03674827
Title: A PHASE 1 STUDY TO EVALUATE THE SAFETY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF ESCALATING DOSES AND TREATMENT INTENSIFICATION OF A VACCINE-BASED IMMUNOTHERAPY REGIMEN-2 (VBIR-2) (PF-06936308) FOR ADVANCED NON-SMALL CELL LUNG CANCER AND METASTATIC TRIPLE-NEGATIVE BREAST CANCER
Brief Title: Vaccine-Based Immunotherapy Regimen For NSCLC and TNBC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to the review of the asset (VBIR-2) within the Sponsor's oncology portfolio; the study was not terminated because of safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C3621001; VBIR-2 (Other: Alias Study Number)
Record Dates: First submitted 2018-08-29; First posted 2018-09-18 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-03

CONDITIONS: Non-Small Cell Lung Cancer; Triple-negative Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Part 1) (Experimental): Participants with NSCLC or TNBC were enrolled at escalating dose levels s of the VBIR-2 regimen.
  Interventions: Biological: PF-06936308
- Dose Expansion (Part 2) (Experimental): Participants with metastatic NSCLC will be enrolled at the expansion dose level identified during Part 1 of the study.
  Interventions: Biological: PF-06936308

INTERVENTIONS:
Biological: PF-06936308 — PF-06936308 components will be administered 4 times per cycle. A cycle is 4 months.
  Other Names: Vaccine-based immunotherapy regimen-2 (VBIR-2)

SUMMARY:
Part 1of the study will evaluate the safety, pharmacokinetics, pharmacodynamics and immunogenicity of increasing doses of a vaccine-based immunotherapy regimen (VBIR-2) for patients with advanced or metastatic non-small cell lung cancer and metastatic triple-negative breast cancer.

Part 2 will evaluate the safety, pharmacokinetics and pharmacodynamics, immunogenicity and preliminary evidence of efficacy of the Expansion dose of VBIR-2 in participants with advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
The study is divided into two parts, Dose Escalation (Part 1) in participants with NSCLC and TNBC without acceptable alternative treatment options, followed by Dose Expansion (Part 2) in participants with NSCLC who have progressed on or after treatment with platinum-based chemotherapy and treatment with 1 immune checkpoint inhibitor, given concurrently or sequentially with chemotherapy.

Part 1 has been completed.

ELIGIBILITY:
Inclusion Criteria:

Part 1:Histological or cytological diagnosis of non-small cell lung cancer or triple-negative breast cancer. Adequate bone marrow, renal and liver function.

Part 2: Histological or cytological diagnosis of metastatic non-small cell lung cancer previously treated with 1 or 2 regimens in metastatic setting including a CPI and platinum-based chemotherapy. Adequate bone marrow, renal and liver function.

Exclusion Criteria:

* Known symptomatic brain metastases
* ECOG performance status greater than or equal to 2
* Concurrent immunotherapy
* History of or active autoimmune disorders (including but not limited to: myasthenia gravis, thyroiditis, pneumonitis, rheumatoid arthritis, multiple sclerosis, systemic lupus, erythematosus, scleroderma) and other conditions that disorganize or alter the immune system.
* History of inflammatory bowel disease.
* Current use of any implanted electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators.
* Presence of any surgical or traumatic metal implants at the site of administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (34):
- United States (34):
  - UCSD Medical Center - Encinitas, Encinitas, California
  - UC San Diego Medical Center - La Jolla (Jacobs Medical Center / Thornton Hospital), La Jolla, California
  - UC San Diego Perlman Medical Offices, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCLA Hematology/Oncology - Parkside, Santa Monica, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - UCSD Medical Center - Vista, Vista, California
  - H Lee Moffitt Cancer Center & Research Institute Inc, Tampa, Florida
  - The University of Chicago Medical Center, CCD - Investigational Drug Service Pharmacy, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - Orland Park - University of Chicago Center for Advanced Care, Orland Park, Illinois
  - Horizon Oncology Research, LLC, Lafayette, Indiana
  - InnerVision Advanced Medical Imaging, Lafayette, Indiana
  - The University of Kansas Cancer Center, Investigational Drug Services, Fairway, Kansas
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute Downtown, Louisville, Kentucky
  - Norton Cancer Institute Pharmacy, Downtown Pharmacy, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - Siteman Cancer Center - St. Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University Infusion Center Pharmacy, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Utah, Huntsman Cancer Hospital, Salt Lake City, Utah
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washington Medical Center - Translational Research Unit (TRU), Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3621001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 55 participants were screened and 36 of them were enrolled and treated in this study.
Groups:
- Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg: Participants with advanced non-small cell lung cancer (NSCLC) or metastatic triple negative breast cancer (mTNBC) in Cohort 1A received 2 repeated cycles of treatment, including AdC68 2x10^11 VP intramuscularly (IM) on Day 1 of Cycles 1 and 2, and pDNA 5 mg IM on Days 29, 57, and 85 of Cycles 1 and 2.
- Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg: Participants with advanced NSCLC or mTNBC in Cohort 2A received 2 repeated cycles of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycles 1 and 2, and pDNA 5 mg IM on Days 29, 57, and 85 of Cycles 1 and 2.
- Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg: Participants with advanced NSCLC or mTNBC in Cohort 3A received 2 repeated cycles of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycles 1 and 2, pDNA 5 mg IM and treme 40 mg subcutaneously (SC) on Days 29, 57, and 85 of Cycles 1 and 2. Treme was administered after AdC68 or pDNA.
- Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg: Participants with advanced NSCLC or mTNBC in Cohort 4A received 2 repeated cycles of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycles 1 and 2; pDNA 5 mg IM, treme 40 mg SC, and sasan 130 mg SC on Days 29, 57, and 85 of Cycles 1 and 2. Sasan was administered after AdC68 or pDNA and after Treme.
- Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg: Participants with advanced NSCLC or mTNBC in Cohort 5A received 2 repeated cycles of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycles 1 and 2; pDNA 5 mg IM, treme 40 mg SC, and sasan 300 mg SC on Days 29, 57, and 85 of Cycles 1 and 2. Sasan was administered after AdC68 or pDNA and after treme.
- Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg: Participants with advanced NSCLC or mTNBC in Cohort 6A received 2 repeated cycles of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycles 1 and 2; pDNA 5 mg IM, treme 80 mg SC, and sasan 300 mg SC on Days 29, 57, and 85 of Cycles 1 and 2. Sasan was administered after AdC68 or pDNA and after treme.
Period: Treatment Phase
Arm/Group | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Started | 3 | 5 | 3 | 4 | 5 | 16
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 5 | 3 | 4 | 5 | 16
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 4 | 3 | 4 | 4 | 9
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Global Deterioration of Health Status | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 1
Period: Long-Term Follow-up Phase
Arm/Group | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Started | 3 | 5 | 3 | 4 | 5 | 16
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 5 | 3 | 4 | 5 | 16
Not completed — Death | 2 | 4 | 2 | 3 | 2 | 6
Not completed — Study Terminated by Sponsor | 0 | 0 | 1 | 1 | 2 | 8
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of one of the components of the regimen.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg | Total
Number analyzed (Participants) | 3 | 5 | 3 | 4 | 5 | 16 | 36
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-44 years | 0 | 0 | 0 | 0 | 1 | 3 | 4
  45-64 years | 2 | 2 | 1 | 4 | 3 | 7 | 19
  ≥65 years | 1 | 3 | 2 | 0 | 1 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 4 | 2 | 11 | 24
  Male | 2 | 2 | 0 | 0 | 3 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 3 | 4 | 5 | 16 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 5 | 3 | 4 | 2 | 15 | 32
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Multiracial | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a clinical investigation where participant administered a product; the event did not need to have a causal relationship with the treatment. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect or considered to be an important medical event. AEs included both SAEs and non-serious AEs.
Time Frame: Baseline up to 6 months after End of Treatment (EOT; 22 months in maximum)
Population: The safety analysis set included all enrolled participants who received at least 1 dose of one of the components of the regimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 3 | 5 | 3 | 4 | 5 | 16
Participants
  Number of participants with all-causality AEs | 3 | 5 | 3 | 4 | 5 | 16
  Number of participants with treatment-related AEs | 1 | 5 | 1 | 4 | 3 | 14
  Number of participants with all-causality SAEs | 2 | 4 | 2 | 3 | 1 | 6
  Number of participants with treatment-related SAEs | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With AEs as Graded by National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE v5.0) (Grade ≥3)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Grades of AEs were defined by NCI CTCAE v5.0. Grade 1 = asymptomatic/mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2 = minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily living (ADL); Grade 3 = severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care ADL; Grade 4 = events with life-threatening consequences, urgent intervention indicated; Grade 5 = death related to AE.
Time Frame: Baseline up to 6 months after EOT (22 months in maximum)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 3 | 5 | 3 | 4 | 5 | 16
Participants
  Grade 3 or Grade 4 (all-causality) | 1 | 1 | 0 | 1 | 2 | 2
  Grade 3 or Grade 4 (treatment-related) | 0 | 0 | 0 | 0 | 1 | 1
  Grade 5 (all-causality) | 2 | 4 | 2 | 1 | 1 | 6
  Grade 5 (treatment-related) | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With AEs Leading to Discontinuation or Dose Reduction
Description: An AE was any untoward medical occurrence in a clinical investigation where participant administered a product; the event did not need to have a causal relationship with the treatment.
Time Frame: Baseline up to 6 months after EOT (22 months in maximum)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 3 | 5 | 3 | 4 | 5 | 16
Participants
  Number of participants with permanent discontinuations | 2 | 0 | 2 | 1 | 1 | 2
  Number of participants with dose reduction or temporary discontinuations | 0 | 0 | 0 | 0 | 2 | 2

4. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: AEs in the first 28 d (days) following the first AdC68 vaccination that were considered possibly related to study treatment and not to disease/progression were DLTs: Grade≥3 neutropenia lasting>7 d, febrile neutropenia, Grade≥3 neutropenic infection, Grade≥3 thrombocytopenia with Grade≥2 clinically significant bleeding, Grade≥3 anemia lasting >7 d, Grade≥3 lymphopenia lasting>14 d; Grade≥3 lab abnormalities associated with symptoms or worsening of an existing condition or that suggested a new disease process or that required additional active management, Grade≥3 AEs considered non-hematologic, non-hepatic major organ toxicity, Grade 3 flu-like symptoms lasting>3 d, fever of >40.0 degree Celsius lasting>3 d, concurrent aspartate aminotransferase or alanine aminotransferase >3x upper limit of normal (ULN) and total bilirubin >2x ULN (potential Hy's law case). Other clinically important or persistent toxicities at discretion of investigator and Pfizer.
Time Frame: The first 28 days following the first AdC68 vaccination (Cycle 1 Day 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 3 | 5 | 3 | 4 | 5 | 16
Participants | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Laboratory Abnormalities in Hematology and Coagulation (Grade 3 or 4)
Description: Laboratory abnormalities (graded per NCI CTCAE v5.0: Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated) in at least 1 participant with data in the categories are presented here. Hematology parameters included hemoglobin, platelets, white blood cell (WBC) count, neutrophils, eosinophils, monocytes, basophils and lymphocytes. Coagulation should include prothrombin time (PT) or international normalized ratio (INR) and activated partial thromboplastin time (APTT).
Time Frame: Baseline up to 6 months after EOT (22 months in maximum)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 3 | 5 | 3 | 4 | 5 | 16
Participants
  APTT prolonged | 0 | 0 | 1 | 1 | 1 | 1
  Anemia | 0 | 0 | 2 | 0 | 0 | 0
  Lymphocyte count decreased | 0 | 0 | 1 | 0 | 0 | 3
  Neutrophil count decreased | 0 | 0 | 0 | 0 | 2 | 0
  Platelet count decreased | 0 | 0 | 1 | 0 | 0 | 0
  WBC count decreased | 0 | 0 | 0 | 0 | 1 | 0

6. Primary Outcome: Number of Participants With Laboratory Abnormalities in Chemistry (Grade 3 or 4)
Description: Chemistry abnormalities (graded per NCI CTCAE v5.0: Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated) in at least 1 participant with data in the categories are presented here. Chemistry parameters included aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, sodium, potassium, magnesium, total chloride, total calcium, total bilirubin, blood urea nitrogen (or urea), creatinine, uric acid, glucose (nonfasted), albumin, phosphorous or phosphate, lactate dehydrogenase, lipase, amylase, bicarbonate or carbon dioxide, total protein, TSH (reflex free T4 and free T3).
Time Frame: Baseline up to 6 months after EOT (22 months in maximum)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 3 | 5 | 3 | 4 | 5 | 16
Participants
  Alanine aminotransferase increased | 0 | 0 | 0 | 0 | 0 | 1
  Alkaline phosphatase increased | 0 | 0 | 0 | 1 | 0 | 0
  Aspartate aminotransferase increased | 0 | 0 | 1 | 1 | 0 | 1
  Blood bilirubin increased | 0 | 0 | 0 | 0 | 0 | 1
  Hyperglycemia | 0 | 1 | 0 | 0 | 2 | 0
  Hyperkalemia | 0 | 1 | 0 | 0 | 0 | 0
  Hyponatremia | 0 | 0 | 1 | 1 | 0 | 1
  Hypophosphatemia | 0 | 2 | 0 | 0 | 0 | 1
  Lipase increased | 0 | 0 | 0 | 1 | 1 | 0
  Serum amylase increased | 0 | 0 | 0 | 1 | 1 | 0

7. Primary Outcome: Number of Participants With Laboratory Abnormalities in Urinalysis (Grade 3 or 4)
Description: Urinalysis abnormalities (graded per NCI CTCAE v5.0: Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated) in at least 1 participant with data in the categories are presented here. Urine parameters included urine protein and urine blood.
Time Frame: Baseline up to 6 months after EOT (22 months in maximum)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 3 | 5 | 3 | 4 | 5 | 16
Participants | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Proportion of Participants Who Achieved Complete Response, Partial Response or Stable Disease for More Than 6 Months Using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Criteria (Part 2)
Description: Clinical Benefit Rate (CBR) is defined as the proportion of participants who achieved anti-tumor responses of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) for >6 months. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). All target lesions must be assessed. PR was defined as ≥30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease and no new lesions. All target lesions must be assessed. SD: Does not qualify for CR, PR or Progression. SD can follow PR only in the rare case that the sum increases by <20% from the nadir, but enough that a previously documented 30% decrease no longer holds.
Time Frame: Performed every 8 weeks from baseline up to Week 32
Population: All enrolled participants who received at least 1 dose of all regimen components administered on Cycle 1 Day 1 and must at least 1 valid and determinate assay result related to the proposed analysis. This was a primary endpoint of Part 2. Part 2 of the study was never opened as the study terminated.
Arm/Group | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Sasanlimab
Description: Cmax was defined as the maximum observed serum concentration.
Time Frame: Cycle 1: at pre-dose on Days 1, 3-6, 8, 15, 22, 29, 57, 85; Cycle 2: at pre-dose on Day 1 and Day 29; EOT; Months 2, 4, and 6 after EOT visit
Population: According to PK analysis reporting defined in protocol, the concentration-time data of sasan after the 1st dose were analyzed individually by noncompartmental methods to determine PK parameters for participants in Cohorts 4A and 5A. Sasan PK parameters in Cohort 6A were not calculated because by design only sparse PK samples were collected. Cohorts 1A, 2A and 3A were not included in the analysis since sasan was not administered in those cohorts.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg
Number analyzed (Participants) | 4 | 4
nanogram per milliliter (ng/mL) | 10520 (46) | 15640 (82)

10. Secondary Outcome: Cmax of Tremelimumab
Description: Cmax was defined as the maximum observed serum concentration.
Time Frame: Cycle 1: at pre-dose on Days 1, 3-6, 8, 15, 22, 29, 57, 85; Cycle 2: at pre-dose on Day 1 and Day 29; EOT; Months 2, 4 and 6 after EOT visit
Population: According to PK analysis reporting defined in protocol, the concentration-time data of treme after the 1st dose were analyzed individually by noncompartmental methods to determine PK parameters for participants in Cohorts 3A and 6A. Treme PK parameters in Cohort 4A and 5A were not calculated because only sparse PK samples were collected. Cohorts 1A and 2A were not included in the analysis since treme was not administered in those cohorts.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 3 | 14
ng/mL | 1692 (47) | 4550 (62)

11. Secondary Outcome: Time to Maximum Concentration (Tmax) of Sasanlimab
Description: Tmax was defined as the time to reach maximum observed serum concentration.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg
Number analyzed (Participants) | 4 | 4
Hour | 165.0 [145 to 167] | 251.5 [69.6 to 499]

12. Secondary Outcome: Tmax of Tremelimumab
Description: Tmax was defined as the time to reach maximum observed serum concentration.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 3 | 14
Hour | 284.0 [163 to 334] | 166.0 [69.5 to 683]

13. Secondary Outcome: Area Under the Curve From Time 0 Extrapolated to Infinity (AUCinf) of Sasanlimab
Description: AUCinf was defined as area under the concentration time curve from time 0 extrapolated to infinity. AUCinf of sasanlimab was not reported due to the limited data points during elimination phase, and the lack of a well-characterized terminal phase. A well-characterized terminal phase was defined as one with at least 3 data points, r^2 ≥0.9, and percent of AUCextrap% ≤20%.
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg
Number analyzed (Participants) | 4 | 4
ng*hr/mL | NA (NA) — AUCinf of sasanlimab was not reported due to the limited data points during elimination phase, and the lack of a well-characterized terminal phase. | NA (NA) — AUCinf of sasanlimab was not reported due to the limited data points during elimination phase, and the lack of a well-characterized terminal phase.

14. Secondary Outcome: AUCinf of Tremelimumab
Description: AUCinf was defined as area under the concentration time curve from time 0 extrapolated to infinity. AUCinf of tremelimumab was not reported due to the limited data points during elimination phase, and the lack of a well-characterized terminal phase. A well-characterized terminal phase was defined as one with at least 3 data points, r^2 ≥0.9, and percent of AUCextrap% ≤20%.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 3 | 14
ng*hr/mL | NA (NA) — AUCinf of tremelimumab was not reported due to the limited data points during elimination phase, and the lack of a well-characterized terminal phase. | NA (NA) — AUCinf of tremelimumab was not reported due to the limited data points during elimination phase, and the lack of a well-characterized terminal phase.

15. Secondary Outcome: Trough Concentrations After Multiple Dosing (Ctrough) of Sasanlimab
Description: Ctrough was defined as the drug concentration observed at the last planned timepoint prior to dosing. Ctrough was not calculated for sasanlimab because trough concentration prior to the fifth dose (on Cycle 2 Day 1) were not collected for any participants in Cohorts 4A or 5A.
Time Frame: Cycle 1: at pre-dose on Days 1, 3-6, 8, 15, 22, 29, 57, 85; Cycle 2: at pre-dose on Day 1 and Day 29; Months 2, 4, 6 after EOT visit
Population: as for outcome 9
Arm/Group | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Ctrough of Tremelimumab
Description: Ctrough was defined as the drug concentration observed at the last planned timepoint prior to dosing.
Time Frame: Cycle 1: at pre-dose on Days 1, 3-6, 8, 15, 22, 29, 57, 85; Cycle 2: at pre-dose on Day 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 1 | 2
ng/mL | NA (NA) — Summary statistics were not computed for PK parameters when fewer than 3 participants had non-missing data. | NA (NA) — Summary statistics were not computed for PK parameters when fewer than 3 participants had non-missing data.

17. Secondary Outcome: Objective Response Rate (ORR) Using RECIST v1.1
Description: ORR was defined as the percentage of participants with best overall response based assessment of CR or PR according to RECIST v1.1. Per RECIST v1.1: CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). All target lesions must be assessed. PR was defined as ≥30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease and no new lesions. All target lesions must be assessed.
Time Frame: Performed every 8 weeks from baseline up to Week 32
Population: All enrolled participants who received at least 1 dose of all regimen components administered on Cycle 1 Day 1 and must at least 1 valid and determinate assay result related to the proposed analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 3 | 5 | 3 | 4 | 5 | 16
Percentage of participants | 0 [0.0 to 70.8] | 0 [0.0 to 52.2] | 0 [0.0 to 70.8] | 0 [0.0 to 60.2] | 0 [0.0 to 52.2] | 0 [0.0 to 20.6]

18. Secondary Outcome: Progression-Free Survival (PFS) Using RECIST v1.1 With NSCLC
Description: PFS was defined as the time from start date to date of first documentation of progression, or death due to any cause. Progression was defined as the appearance of local, regional or distant disease of the same type after complete response or progression of pre-existing lesions.
Time Frame: Performed every 3 weeks after treatment discontinuation until death, participant refusal, or lost to follow-up (telephone contact acceptable).
Population: All enrolled participants with NSCLC who received at least 1 dose of all regimen components administered on Cycle 1 Day 1 and must at least 1 valid and determinate assay result related to the proposed analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 3 | 4 | 3 | 9
Months | 2.0 [0.4 to 2.0] | 1.8 [1.8 to 5.3] | 1.8 [1.7 to 1.9] | 1.8 [0.6 to NA] — Not estimable based on the Brookmeyer and Crowley method.

19. Secondary Outcome: PFS Using RECIST v1.1 With TNBC
Description: PFS was defined as the time from start date to date of first documentation of progression, or death due to any cause. Progression was defined as the appearance of local, regional or distant disease of the same type after complete response or progression of pre existing lesions.
Time Frame: as for outcome 18
Population: All enrolled participants with TNBC who received at least 1 dose of all regimen components administered on Cycle 1 Day 1 and must at least 1 valid and determinate assay result related to the proposed analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 1 | 3 | 4 | 2 | 7
Months | 1.2 [NA to NA] — Not estimable based on the Brookmeyer and Crowley method. | 7.0 [2.0 to 12.0] | 1.3 [1.2 to 1.7] | 1.9 [1.7 to 2.0] | 1.8 [0.8 to 3.7]

20. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Against Sasanlimab
Description: Participants were considered ADA-positive if (1) baseline titer was missing or negative and participant had ≥1 post-treatment positive titer (treatment-induced), or (2) positive titer at baseline and had a ratio of ≥4 in titer (dilution) to baseline in ≥1 post-treatment sample (treatment-boosted).
Time Frame: Cycle 1: on Day 1, Day 29, and Day 85; Cycle 2: on Day 29; at the EOT visit, and 2, 4 and 6 months after EOT. Samples to be collected on dosing days were obtained within 6 hours prior to sasanlimab dosing.
Population: All enrolled participants who received at least 1 dose of the VBIR-2 component was the participant of the immunogenicity assessment (tremelimumab or sasanlimab). For this outcome measure, participants who received sasanlimab in Cohorts 4A, 5A and 6A were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 4 | 5 | 16
Participants
  Treatment-induced | 0 | 0 | 0
  Treatment-boosted | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Neutralizing Antibody (NAb) Against Sasanlimab
Description: A participant was NAb positive if (1) baseline titer was missing or negative and participant had ≥1 post-treatment positive titer (treatment-induced), or (2) positive titer at baseline and had a ratio of ≥4 in titer (dilution) to baseline in ≥1 post-treatment sample (treatment-boosted). Participants who were either (1) an ADA-negative participant or (2) an ADA-positive participant without treatment-induced or treatment-boosted NAb response were considered as NAb negative.
Time Frame: as for outcome 20
Population: All enrolled participants who received at least 1 dose of all assigned regimen components administered, and must have had at least 1 valid and determinate assay result related to the proposed analysis. For this outcome measure, NAb against sasanlimab was examined for the 2 participants with ADA positive samples at baseline in Cohort 6A.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 0 | 0 | 2
Participants |  |  | 0

22. Secondary Outcome: Number of Participants With ADA Against Tremelimumab
Description: as for outcome 20
Time Frame: Cycle 1: on Day 1, Day 29, and Day 85; Cycle 2: on Day 29; at the EOT visit, and 2, 4 and 6 months after EOT. Samples collected on dosing days were obtained within 6 hours prior to tremelimumab dosing.
Population: All enrolled participants who received at least 1 dose of the VBIR-2 component was the participant of the immunogenicity assessment (tremelimumab or sasanlimab). For this outcome measure, participants who received tremelimumab in Cohorts 3A, 4A, 5A and 6A were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 3 | 4 | 5 | 16
Participants
  Treatment-induced | 0 | 0 | 0 | 1
  Treatment-boosted | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With NAb Against Tremelimumab
Description: A participant was NAb positive if (1) baseline titer was missing or negative and participant had ≥1 post-treatment positive titer (treatment-induced), or (2) positive titer at baseline and had a ratio of ≥4 in titer (dilution) to baseline in ≥1 post-treatment sample (treatment-boosted). Participants who were either (1) an ADA-negative participant or (2) an ADA-positive participant without treatment-induced or treatment-boosted NAb response were considered as NAb negative. NAb evaluation was not considered as meaningful taken that treatment-induced ADA was found in only 1 participant. Thus, NAb to tremelimumab was not examined.
Time Frame: Cycle 1: on Day 1, Day 29, and Day 85; Cycle 2: on Day 29; at the EOT visit, and 2, 4 and 6 months after EOT. Samples to be collected on dosing days were obtained within 6 hours prior to tremelimumab dosing.
Population: All enrolled participants who received at least 1 dose of all assigned regimen components administered, and must have had at least 1 valid and determinate assay result related to the proposed analysis.
Arm/Group | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

24. Secondary Outcome: Titers of Treatment-Induced ADA and NAb Against Sasanlimab
Description: Titers were measured in terms of 1/dilution. Only the samples tested positive for ADA were to be further tested for Nab. Treatment-induced ADA: baseline titer is missing or negative and participant has >= 1 post-treatment positive titer. Treatment-induced NAb: baseline titer was missing or negative and participant had ≥1 post-treatment positive titer.
Time Frame: Cycle 1: at Day 1, Day 29, and Day 85; Cycle 2: at Day 29; at the EOT visit, and 2, 4 and 6 months after EOT. Samples to be collected on dosing days were obtained within 6 hours prior to sasanlimab dosing.
Population: All enrolled participants who received at least 1 dose of all assigned regimen components administered, and must have had at least 1 valid and determinate assay result related to the proposed analysis. For this outcome measure, participants who received sasanlimab in Cohorts 4A, 5A and 6A were included. No participants had treatment-induced ADA.
Arm/Group | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 0 | 0 | 0

25. Secondary Outcome: Titers of Treatment-Induced ADA and NAb Against Tremelimumab
Description: Titers were measured in terms of 1/dilution. Only the samples tested positive for ADA were to be further tested for Nab. Treatment-induced ADA: baseline titer is missing or negative and participant has >= 1 post-treatment positive titer. Treatment-induced NAb: baseline titer was missing or negative and participant had ≥1 post-treatment positive titer. NAb was not examined as the evaluation was not meaningful considering only 1 participant had treatment-induced ADA.
Time Frame: Cycle 1: at Day 1, Day 29, and Day 85; Cycle 2: at Day 29; at the EOT visit, and 2, 4 and 6 months after EOT. Samples to be collected on dosing days were obtained within 6 hours prior to tremelimumab dosing.
Population: as for outcome 23
Measure: Median (Inter-Quartile Range); unit: 1/dilution
Groups:
- Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg: Participants with advanced NSCLC or mTNBC in Cohort 3A received 2 repeated cycles of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycles 1 and 2, pDNA 5 mg IM and treme 40 mg subcutaneously (SC) on Day 29, 57, and 85 of Cycles 1 and 2. treme were administered after AdC68 or pDNA.
Arm/Group | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
Number analyzed (Participants) | 0 | 0 | 0 | 1
1/dilution
  ADA Titer |  |  |  | NA [NA to NA] — No summary statistics were provided for N <3 considering the insufficient number of participants with event (only 1 participant with treatment-induced ADA).
  NAb Titer: number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 6 months after EOT (22 months in maximum)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. AE reporting, including suspected unexpected serious adverse reactions, was carried out in accordance with applicable local regulations.
Arm/Group | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/5 | 2/3 | 3/4 | 2/5 | 6/16
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/5 | 2/3 | 3/4 | 1/5 | 6/16
Other Adverse Events (participants affected / at risk) | 2/3 | 5/5 | 3/3 | 4/4 | 5/5 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg (N=3) | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg (N=5) | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg (N=3) | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg (N=4) | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg (N=5) | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg (N=16)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Renal vein thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1A Adenovirus C68 (AdC68) 2X10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg (N=3) | Cohort 2A AdC68 6X10^11 VP + pDNA 5 mg (N=5) | Cohort 3A AdC68 6X10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 40 mg (N=3) | Cohort 4A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasanlimab (Sasan) 130 mg (N=4) | Cohort 5A AdC68 6X10^11 VP + pDNA 5 mg + Treme 40 mg + Sasan 300 mg (N=5) | Cohort 6A AdC68 6X10^11 VP + pDNA 5 mg + Treme 80 mg + Sasan 300 mg (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (4) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 5 (6)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 6 (6)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 3 (4) | 7 (10)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 3 (3)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (8)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 3 (8)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electric shock sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Penile rash (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 5 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated on 10 Feb 2021 by the Sponsor. The decision to terminate this study was based on the results of a strategic evaluation of VBIR-2 within the current Sponsor's oncology portfolio. When the decision of study termination was made, participants enrolled in Part 1 who were still on study were to remain on treatment until 31 Aug 2021; Part 2 of the study was never opened.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT03674827/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT03674827/SAP_001.pdf